CLINICAL TRIAL: NCT00530478
Title: Effect of Donepezil on the Reorganization of Cognitive Neural Network in Patients With Post-Stroke Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2006-04-023
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2007-07

CONDITIONS: Stroke
Keywords: Donepezil; Stroke; Cognitive function; Cognitive neural network
MeSH Terms: conditions — Stroke | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Donepezil

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of donepezil on the recovery of cognitive function in patients with stroke and to delineate the neurophysiologic mechanisms of the therapeutic effect of donepezil on the recovery of cognitive network using functional neuroimaging technique.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke in the territory of right or left middle cerebral artery
* Post-onset duration of the recent-onset stroke is over 3 months
* Cognitive deficit ranged from 10 to 26 by minimal mental status examination (MMSE) score
* Disturbance in activities of daily living (ADL) ranged 0.5 ~ 2.0 by clinical dementia rating (CDR) scale

Exclusion Criteria:

* Severe internal carotid artery stenosis on the lesion side
* Cardiac pacemaker or intracranial metal insertion
* Post-stroke seizure disorder or any evidence of epileptic spikes on electroencephalography (EEG)

Ages: 16 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Suk Hoon Ohn, MD, MS, Principal Investigator — Samsung Medical Center; Yun Hee Park, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea